CLINICAL TRIAL: NCT03675412
Title: Acute Changes in Optic Nerve Head (ONH) and Macular Blood Flow After Caffeine Consumption in Glaucoma Patients and Healthy Subjects: A Quantitative Optic Coherence Tomography Angiography (OCTA) Study
Brief Title: Caffeine Consumption in Glaucoma Patients and Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, M. Reza Razeghinejad MD, Principal Investigator, Wills Eye
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB#18-729
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma, Primary Open Angle
Keywords: Primary Open Angle Glaucoma (POAG); Optical Coherence Tomography Angiography (OCTA); Caffeine; Macular Blood Flow; Peripapillary Blood Flow
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: All eyes will undergo imaging to measure blood flow in the back of the eye (retina and optic nerve) using the Avanti AngioVue HD OCTA (optical coherence tomography angiography)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glaucoma Patients (Active Comparator): Eligible participants include patients with mild, moderate or advanced primary open angle glaucoma (POAG) or primary angle closure glaucoma (PACG). Each participant will complete baseline study tasks. Each participant will then receive one 200 mg caffeine tablet to ingest. Study tasks will be performed 1 hour and 2 hours after caffeine ingestion.
  Interventions: Dietary Supplement: Caffeine tablet
- Healthy controls (Active Comparator): Eligible participants include healthy subjects with no eye diseases. Each participant will complete baseline study tasks. Each participant will then receive one 200 mg caffeine tablet to ingest. Study tasks will be performed 1 hour and 2 hours after caffeine ingestion.
  Interventions: Dietary Supplement: Caffeine tablet

INTERVENTIONS:
Dietary Supplement: Caffeine tablet — Each eligible participant will receive one 200 mg caffeine tablet to ingest after completing all baseline study tasks.

SUMMARY:
Caffeine is the most widely consumed drinking nutrient in the world. Caffeine effects various organs and the vascular system. It decreases ocular blood flow due to vasoconstriction.

DETAILED DESCRIPTION:
Ingestion of caffeine in glaucoma patients and healthy subjects may decrease peripapillary and macular blood flow in the back of the eye.

The primary objective of this study is to assess the acute changes in peripapillary and macular blood flow before and after an intake of oral caffeine (200 milligram tablet) in glaucoma patients and healthy subjects by using optical coherence tomography angiography (OCTA) scans. This novel imaging tool creates three-dimensional angiograms to assesses signal changes caused by flowing blood cells in a non-invasive angiogram scan. Blood flow is shown as vessel density measured in percentage.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 90 years
* diagnosis of primary open angle glaucoma (Mild, Moderate and Advanced)
* healthy subjects with no eye disease

Exclusion Criteria:

* Diseases, ophthalmic or systemic, that are likely to affect OCTA results
* greater than moderate cataract
* nystagmus
* inability to look at target
* macular degeneration other than mild drusen or pigmentary changes
* diabetic retinopathy
* neovascular glaucoma or non-glaucoma optic neuropathies
* current macular edema, prior laser to retina, inflammatory retinopathy or choroidopathy
* keratoconus, corneal ectasia, central corneal scarring
* rheumatologic diseases or Raynaud's phenomena
* pregnant and lactating women
* mental illness or alcohol addiction
* pre-existing bladder symptoms, cardiac disease or sleep disorder
* refractive spherical diopter greater than 5 or cylinder greater than 3
* possible tolerance to caffeine (drinking more than 1 cup coffee per day).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow change in back of eye before and after caffeine | Baseline, Hour 1, Hour 2
  Optical Coherence Tomography Angiography (OCTA) will be obtained using the Avanti AngioVue High Definition (HD) OCTA by Optovue. Images will include standard 4.5mm HD disc scan, 6mm HD retina scan, regular optic nerve head (ONH) structural scan, 3D-disc baseline scan and a regular ganglion cell complex analysis (GCCA) structural scan. This will measure blood flow changes in the back of the eye by imaging vessel density in percentage before then 1 and 2 hours after caffeine.

CONTACTS AND LOCATIONS:
Overall Officials: M. Reza Razeghinejad, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03675412/Prot_000.pdf